CLINICAL TRIAL: NCT05705739
Title: Comparison Between the Efficacy of Ultrasound Guided Erector Spinae Plane Block Versus Retrolaminar Plane Block for Postoperative Pain in Patients Undergoing Hepatobiliary Surgery
Brief Title: Ultrasound Guided Erector Spinae Plane Block Versus Retrolaminar Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Hassan Mokhtar Elshorbagy Hetta, lecturer of anesthesia and ICU, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 544/2022
Record Dates: First submitted 2023-01-20; First posted 2023-01-31 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Post Operative Pain; Analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retrolaminar plane block (Experimental)
  Interventions: Procedure: retrolaminar block
- ESPB (Experimental)
  Interventions: Procedure: ESPB

INTERVENTIONS:
Procedure: retrolaminar block — curved probe will be placed 1-1.5 cm lateral to the target spinous process after identification of the lamina, the needle will be advanced caudally until it contacts the lamina
  Arms: Retrolaminar plane block
Procedure: ESPB — curved probe will be placed 2-3 cm lateral to the spine using a sagittal approach at the level of T8. After identification of erector spinae muscle and transverse processes, the needle will be inserted deeply into the erector spinae muscle.
  Arms: ESPB

SUMMARY:
Retrolaminar block (RLB) and erector spinae plane block (ESPB) are alternative approaches to paravertebral block (PVB) and are advantageous in that they are easier and safer techniques compared with the traditional PVB. These blocks are considered to be compartment blocks or interfascial plane blocks. In these approaches, local anesthetics are assumed to penetrate the superior costotransverse ligament and reach the paravertebral space, although the needle tip is not advanced into the paravertebral space.

the study aim to evaluate and compare the analgesic efficacy of retrolaminar plane block and erector spinae plane block.

ELIGIBILITY:
Inclusion Criteria:

1. Age18-60.
2. Both genders.
3. hepatobiliary surgery.
4. ASA I-III.

Exclusion Criteria:

1. Drug allergy.
2. Morbid obesity (BMI >40 kg/m2).
3. Psychiatric disorder.
4. Opiod dependence.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Visual analogue pain scale | 24 hour
  score from 0-10 (0 mean no pain and 10 the worst pain )

SECONDARY OUTCOMES:
Time of first post operative analgesic request. | 24 hour
  time to demand rescue analgesia
Total analgesic consumption | 24 hour
  total fentanyl consumption during the first day postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No